CLINICAL TRIAL: NCT01504230
Title: Multi-joint Coordination Underlies Upright Balance Control in Elderly With Osteoporosis
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201104056RB
Record Dates: First submitted 2012-01-03; First posted 2012-01-05 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Osteoporosis
Keywords: To ascertain the mechanisms for effectively controlling balance in seniors with osteoporosis and to provide a basis for developing fall prevention programs.; To develop biomechanical models that control the entire body's center of mass (CoM) during upright quiet stance in seniors with osteoporosis.; To identify the mechanism to control the entire body's CoM after receiving a balance perturbation in seniors with osteoporosis.
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- health older adults
- Osteoporosis participants

SUMMARY:
Osteoporosis is a prevalent health concern among older adults and is associated with an increased risk of falls that can cause fracture, injury and even mortality. Identifying the factors related to falls occur within this population is essential for the development of effective regimes for fall prevention. The long-term objectives of this work are to ascertain the mechanisms for effectively controlling balance in seniors with osteoporosis and to provide a basis for developing fall prevention programs. The entire body's center of mass (CoM) is a critical indicator for balance control and the coordination among joints and muscles to control the CoM is still unclear. The aim1 of this study is to develop biomechanical models that control the entire body's center of mass (CoM) during upright quiet stance in seniors with osteoporosis. The aim2 of this study is to identify the mechanism to control the entire body's CoM after receiving a balance perturbation in seniors with osteoporosis. The findings of this research can provide needed information regarding the processes of balance control in this vulnerable osteoporosis population, and has the potential to be applied to individuals with other neuromuscular and orthopedic deficits.

ELIGIBILITY:
Inclusion Criteria:

* for healthy older adults (OA)

  1. can stand for 5 minutes and walk for 6 minutes independently
  2. normal or corrected to normal vision
  3. an age between 65-85 years
  4. no osteoporosis (T-score above -2.5)
* for osteoporosis participants (OP)

  1. can stand for 5 minutes and walk for 6 minutes independently
  2. normal or corrected to normal vision
  3. an age between 65-85 years
  4. no osteoporosis (T-score below -2.5)

Exclusion Criteria:

1. pregnant women
2. cancer diagnosis
3. sensory-motor deficits
4. the BMI is larger than 30 or smaller than 18

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Hsu, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- School & Graduate Institute of Physical Therapy College of Medicine, National Taiwan University, Taipei, Taiwan